CLINICAL TRIAL: NCT04158271
Title: Evaluation of Techniques for Tracheal Tube Exchange in Standard and Critical Care Patients
Acronym: TUBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUU
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Airway Morbidity
Keywords: Airway Management; Tube Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prone Position (Experimental): Evaluation of Techniques for tracheal tube Exchange in prone position
  Interventions: Device: Prone Position; Device: Laryngeal tube; Device: Endotracheal tube Leackage
- Laryngeal tube (Experimental): Evaluation of Techniques for tracheal tube Exchange in patients with laryngeal tube (LT)
  Interventions: Device: Prone Position; Device: Laryngeal tube; Device: Endotracheal tube Leackage
- Endotracheal tube Leackage (Experimental): Evaluation of Techniques for tracheal tube Exchange in critical care patients with a endotracheal tube and a high leackage
  Interventions: Device: Prone Position; Device: Laryngeal tube; Device: Endotracheal tube Leackage

INTERVENTIONS:
Device: Prone Position — In a randomized order we evaluate techniques for securing the airway in paralyzed patients in prone position
Device: Laryngeal tube — In a randomized order we evaluate techniques for securing the airway in patients with a failed laryngeal tube
Device: Endotracheal tube Leackage — In a randomized order we evaluate techniques for securing the airway in paralyzed patients with a endotracheal tube and a cuff leackage

SUMMARY:
A randomized controlled study to evaluate different Techniques and Approachs for the Exchange of a tracheal tube or supraglottic airway device in a Simulator

DETAILED DESCRIPTION:
Exchanging a tracheal tube (ETT) in the high-risk difficult airway patient carries the risk of hypoxemia and the potential of a lost airway. Maintaining continuous airway access during the exchange by incorporating an airway exchange catheter (AEC) or similar device may reliably lessen exchange risk, especially in the known or suspected difficult airway patient, by providing a conduit to facilitate ETT passage into the trachea. We evaluated some approven / etablished techniques in a Simulator based study design.

ELIGIBILITY:
Inclusion Criteria:

* residents and consultans of the Department of Anesthesiology

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of Strategies for Securing the Airway | through study completion, an average of 10 minutes
  Evaluation of Strategies for securing the Airway in patients in the OR and Critical Care Medicine. Participants are confronted with three airway scenarios and perform in a Simulator different airway management strategies.

SECONDARY OUTCOMES:
Time for intervention | through study completion, an average of 10 minutes
  time for Exchange the Primary airway device
Anaesthesia Experience | through study completion, an average of 10 minutes
  individual anaesthesia experience
IDS | through study completion, an average of 10 minutes
  after the Scenario we calculate the Intubation difficult score (IDS)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Center of Johannes Gutenberg-University
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany